CLINICAL TRIAL: NCT03281486
Title: Clinical Evaluation of the Efficacy of "Hyaluronan" Formulation for Dry Mouth in Patients With Type 2 Diabetes
Brief Title: "Hyaluronan" Formulation for Type 2 Diabetic Patients With Dry Mouth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: You First Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LUD-105-17
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Dry Mouth; Xerostomia; Type 2 Diabetics
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HA formulation Oral Spray (Experimental): Subjects will be instructed to mouth spray with 0.3 ml ( 2 sprays to the mouth) of their assigned mouth spray, 2 times daily (morning and evening), using only the assigned mouth spray provided for the 4 week duration of the study.
  Interventions: Device: HA formulation Oral Spray
- Placebo Oral Spray (Placebo Comparator): Subjects will be instructed to mouth spray with 0.3 ml ( 2 sprays to the mouth) of their assigned mouth spray, 2 times daily (morning and evening), using only the assigned mouth spray provided for the 4 week duration of the study.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: HA formulation Oral Spray — It is an HA formulation of FDA listed ingredients
  Arms: HA formulation Oral Spray
Device: Placebo — Placebo formulation without the active ingredients
  Arms: Placebo Oral Spray

SUMMARY:
An increased incidence of dental caries in association with poorly controlled diabetes has also been reported, Xerostomia (dry mouth) has been reported to be a common complaint of patients with diabetes, Without adequate saliva production, both hard and soft tissues of the mouth can be severely damaged and become more susceptible to infections. This 9 week, cross-over group, randomized, single center, study will evaluate the efficacy of HA formulation in alleviating dry mouth in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient should be above 18 years of age.
2. Patients who have been diagnosed with type 2 diabetes and have developed dry mouth or have worsening of pre-existing dry mouth condition.
3. Ability to attend visits at the research site
4. Patient should be able to read and/or understand and sign the consent form and be willing to participate in the research study
5. Agree to abstain from the use of any products for xerostomia other than those provided in the study.
6. Agree to comply with the conditions and schedule of the study.

Exclusion Criteria:

1. Subjects with open mouth sores at study entry.
2. Any pathology that, based on the judgement of the researcher, could negatively affect the oral mucosa and subsequent treatment for xerostomia.
3. Subjects who are nursing, becoming pregnant or plan to become pregnant during the study period
4. Subjects currently on medication or treatment for dry mouth/xerostomia
5. Hypersensitivity to any of the following ingredients- HA ,xylitol and Sodium Benzoate.
6. Subjects with soft or hard tissue tumor of the oral cavity.
7. Presence of severe gingivitis.
8. Chronic disease with concomitant oral manifestations other than xerostomia
9. History of radiation therapy to head and neck
10. Subjects with conditions the investigator may feel will interfere with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Relief from drymouth using VAS scoring | 9 weeks
  Patients' perception of efficacy of a new mouth spray for 9 weeks in reducing the symptoms of drymouth in diabetic patients using VAS scoring

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology and Metabolism, Saint Louis University, St Louis, Missouri, United States